CLINICAL TRIAL: NCT00947674
Title: Prospective, Randomized, Double-Blind, Sham Treatment Controlled Multicenter Study to Evaluate Efficacy and Safety of Cellsorba™EX Used for Leukocytapheresis (LCAP) in Patients With Steroid-Free, Active Ulcerative Colitis
Brief Title: A Study of Leukocytapheresis (LCAP) in Patients With Ulcerative Colitis (UC)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: short of enrollment
Sponsor: Asahi Kasei Medical Co., Ltd. (Industry)
Collaborators: Asahi Kasei Medical Europe GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEWS80
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Ulcerative Colitis
Keywords: Cellsorba EX
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cellsorba EX (Experimental)
  Interventions: Device: Cellsorba EX
- Sham treatment (Sham Comparator)
  Interventions: Device: Cellsorba EX

INTERVENTIONS:
Device: Cellsorba EX — conduct treatment twice a week for 3 weeks and once a week for 4 weeks, total 10 times

SUMMARY:
This is a prospective, randomized, double-blind, sham treatment controlled multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed to have UC in the active stage based on clinical symptoms and findings from endoscopy
* Patients with pancolitis type or left-sided colitis type lesion of 15 cm or longer observed endoscopically
* Patients with Mayo score between 5 and 10
* Patients with Mayo sub-score (findings from flexible sigmoidoscopy) of 2 or 3
* Patients not having received any corticosteroids (referred to as steroids) (p.o., i.v., enema, suppository) within the past 6 weeks

Exclusion Criteria:

* Patients with a difficulty in peripheral vascular access
* Patients having received ACE inhibitor (at least 10 times of its half-life time for interval needed before initiating the treatment)
* Patients with toxic megacolon
* Patients with a malignant disease or its experience
* Patients with a severe cardiovascular disease (grade III or IV by the Classification of heart functions of the New York Heart Association (NYHA))
* Patients with a liver or kidney disease (AST(GOT) or ALT(GPT) or total bilirubin or creatinine level which is 2 or more times higher than the upper limit of normal (abbreviated as ULN, hereinafter)
* Patients suspected to have or having HBV or HCV or HIV or pathogenic bacteria
* Patients on anticoagulant therapy or with abnormality in the blood coagulation system (PT or PTT levels which are 1.5 or more times higher than ULN
* Pregnant women or patients with possible pregnancy
* Breast feeding women
* Patients weighing 40 kg or less
* Patients with hemoglobin level of less than 6.5 mmol/L (10.5 g/dL)
* Patients with platelet count of less than 150 x 103/mm3, 150 x 109/L (15 x 104/mm3)
* Patients with white blood cell count of less than 3.5 x 109/L (3,500/mm3)
* Patients with hypotension (with systolic blood pressure of 80 mmHg or less)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-05; Primary Completion 2012-01 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Clinical response | at 8th week

SECONDARY OUTCOMES:
Remission, Mayo scores, Mucosal healing, CRP | at 8th and 16th week

CONTACTS AND LOCATIONS:
Locations (10):
- Prague, Czechia
- Germany (2):
  - Hanover
  - Rostock
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Japan (2):
  - Hyōgo
  - Tokyo
- Sweden (2):
  - Gothenburg
  - Stockholm
- United Kingdom (2):
  - Oxford
  - Southampton